CLINICAL TRIAL: NCT02084433
Title: Comparison of Intraosseous Anaesthesia Using a Computerized System (QuickSleeper) to Conventional Anesthesia
Acronym: QUICK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Frederic COURSON, assistant professor, hospital practitionner, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75018
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Deep Caries; Molar Incisor Hypomineralisation
Keywords: MIH of the first permanent molar
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional anasthesia (Active Comparator): para-apical maxillary and locoregional mandibular (Articaine 1/100000) anaesthesia
  Interventions: Procedure: conventional anasthesia
- intraosseous anaesthesia (Experimental): intraosseous anaesthesia using a computerized system (Quicksleeper) "1 / Anesthesia of periosteum (Articaine 1/100000) 2 / penetration of the needle rotated to the apex 3 / osteocentral injection "
  Interventions: Procedure: intraosseous anaesthesia using a computerized system

INTERVENTIONS:
Procedure: intraosseous anaesthesia using a computerized system — "1 / Anesthesia of periosteum (Articaine 1/100000) 2 / penetration of the needle rotated to the apex 3 / osteocentral injection "
  Arms: intraosseous anaesthesia
Procedure: conventional anasthesia — para-apical maxillary and locoregional mandibular (Articaine 1/100000) anaesthesia
  Arms: conventional anasthesia

SUMMARY:
The purpose is to compare the efficacy of an intraosseous anaesthesia using a computerized system (QuickSleeper) to a conventional infiltration anesthesia. Our hypothesis is that anesthesia via QuickSleeper system can reduce pain during anesthesia and obtain a more rapid local anesthesia compared to the anesthesia via conventional technique by infiltration.

Design: split-mouth design AND parallel-arm design

DETAILED DESCRIPTION:
Local anesthesia is commonly used in oral health care and intra-mucosal infiltration anesthesia is most commonly used by practitioners. Anesthesia may cause children a great deal of anxiety because of the fear of the injection. The latter can be painful if the product is delivered too quickly in the mucosa. Recent developments in the techniques and anesthesia systems allow reducing pain during the injection. In particular, computerized systems (electronically assisted local anesthesia) allow a slow injection limiting pressure. Moreover, these systems look like a pen which prevents the negative impression of the image related to the syringe metal. The intraosseous electronically-assisted anesthesia could be an interesting alternative to conventional infiltration anesthesia by making the act less stressful but also less painful for the child.

ELIGIBILITY:
Inclusion Criteria:

* split-mouth randomized controlled trial: patients with at least two first permanent molars requiring the same treatment with anesthesia
* parallel-arm radnomized controlled trial: patients with first permanent molar requiring treatment with anesthesia
* vital pulp
* patient did not take any pain medication 48 hours before randomization
* non-opposition of the child and two holders of parental participation in the study
* Treatments can be conservative treatment or endodontic treatment limited to pulpotomy.

Exclusion Criteria:

* Patients with periodontal disease (periodontal pockets or tooth mobility) or radiological defects (necrosis, furcation or periapical radiolucency)
* Disabled or autistic patients
* Patients with cancer, heart disease or sickle cell anemia

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pain reported by the patient according to the visual analogue scale (VAS) | up to 10 minutes
  Pain reported by the patient according to the visual analogue scale (VAS) will be evaluated at the end of the injection / infiltration. The assessment will concern the insertion of the needle and the injection / infiltration

SECONDARY OUTCOMES:
latency | up to 15 minutes
  latency (in minutes) evaluated by examining the sensitivity of the sulcus using a probe (an exam will be conducted every minute until the sulcus is insensitive to the probe)
need for additional anesthesia during the treatment | 1 hour
pain felt during the treatment | 1 hour
  need for additional anesthesia during the treatment; pain felt during the treatment evaluated at the end of treatment according to the VAS

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Courson, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France

REFERENCES:
- [Derived] Smail-Faugeron V, Muller-Bolla M, Sixou JL, Courson F. Evaluation of intraosseous computerized injection system (QuickSleeper) vs conventional infiltration anaesthesia in paediatric oral health care: A multicentre, single-blind, combined split-mouth and parallel-arm randomized controlled trial. Int J Paediatr Dent. 2019 Sep;29(5):573-584. doi: 10.1111/ipd.12494. Epub 2019 Apr 8. PMID 30883951
- [Derived] Smail-Faugeron V, Muller-Bolla M, Sixou JL, Courson F. Split-mouth and parallel-arm trials to compare pain with intraosseous anaesthesia delivered by the computerised Quicksleeper system and conventional infiltration anaesthesia in paediatric oral healthcare: protocol for a randomised controlled trial. BMJ Open. 2015 Jul 10;5(7):e007724. doi: 10.1136/bmjopen-2015-007724. PMID 26163031